CLINICAL TRIAL: NCT06252792
Title: Prospective, Multicenter, Open and Non-interference Observational Clinical Study of Daratumumab, Pomalidomide and Dexamethasone (Dara-PD) in the Treatment of Patients With First Relapse of Multiple Myeloma
Brief Title: Dara-PD in the Treatment of Patients With First Relapse of Multiple Myeloma
Status: Not yet recruiting | Type: Observational
Sponsor: FengYan Jin (Other)
Collaborators: Affiliated Hospital of Hebei University (Other); Second Hospital of Shanxi Medical University (Other); Shandong Cancer Hospital and Institute (Other); First Affiliated Hospital of Jinan University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, FengYan Jin, Clinical Professor of Hematology Department, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: First relapse multiple myeloma
Record Dates: First submitted 2023-12-21; First posted 2024-02-12 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma; First Relapse
Keywords: Multiple Myeloma; First relapse; the second progression free survival time (PFS2)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood、bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- daratumumab, pomalidomide, and dexamethasone (Dara-PD): the first relapse of patients who received daratumumab, pomalidomide, and dexamethasone (Dara-PD) treatment
- other regimens in the same period (including Dara-KPD, VPd, KPd, IPd, Pd): the first relapse of patients who received other regimens in the same period (including Dara-KPD, VPd, KPd, IPd, Pd) treatment

SUMMARY:
At present, there is no prospective study on the treatment of first-relapsed multiple myeloma with daratumumab plus pomalidomide and dexamethasone (Dara-Pd). A prospective, multicenter, open, non-interventional, observational clinical study to evaluate the efficacy and safety of Dara-Pd in patients with first relapse multiple myeloma.

DETAILED DESCRIPTION:
To evaluate the impact of daratumumab, pomalidomide, and dexamethasone (Dara-PD) compared to other regimens in the same period (including Dara-KPD, VPd, KPd, IPd, Pd) on the second progression free survival time (PFS2) of first relapse of multiple myeloma. Among them, the second progression free survival time (PFS2) is defined as the time from enrollment to disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled in this study only if they met all of the following inclusion criteria.

1. Age 18 years or older, regardless of gender.
2. Diagnosis of symptomatic multiple myeloma based on the 2014 IMWG diagnostic criteria and the presence of measurable disease
3. First relapse of multiple myeloma;
4. Receiving first-line anti-multiple myeloma therapy;
5. The first-line therapy must be based on proteasome inhibitors and immunomodulators (RVD);
6. Subject must have achieved a response (partial response [PR] or better based on investigator's determination of response by the IMWG criteria) to at one prior regimen;
7. Each subject (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.
8. Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. Contraception must begin 4 weeks prior to dosing and continue until at least 3 months after receiving the last dose of the study drug. A woman of childbearing potential must have a negative serum or urine pregnancy tests at screening within 14 days prior to randomization.

Exclusion Criteria:

1. Diagnosis of inactive multiple myeloma, including primary amyloidosis, MGUS (monoclonal gammopathy of undetermined significance) or smoldering myeloma.
2. Relapsed and refractory myeloma：Relapsed and refractory myeloma is defined as disease that is nonresponsive while on salvage therapy, or progresses within 60 days of last therapy in patients who have achieved minimal response (MR) or better at some point previously before then progressing in their disease course；
3. Primary refractory myeloma：Primary refractory myeloma is defined as disease that is nonresponsive in patients who have never achieved a minimal response or better with any therapy；
4. Subject has received daratumumab or pomalidomide previously；
5. Subject has a history of malignancy (other than multiple myeloma) within 3 years before the date of randomization (exceptions is malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years).；
6. Subjects with uncontrollable psychiatric disorders;
7. Subject is known or suspected of not being able to comply with the study protocol.Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the first relapse of multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
the second progression free survival time (PFS2) | through study completion, up to 2 years
  daratumumab, pomalidomide, and dexamethasone (Dara-PD) compared to other regimens in the same period (including Dara-KPD, VPd, KPd, IPd, Pd) on the second progression free survival time (PFS2) of first relapse of multiple myeloma.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | through study completion, up to 2 years
  Evaluated according to the 2016 IMWG efficacy evaluation criteria, defined as the proportion of participants who achieved the best response as strict complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
Deep response rate (≥ VGPR) | through study completion, up to 2 years
  Evaluated according to the 2016 IMWG efficacy evaluation criteria, defined as the proportion of subjects who achieved the best response as strict complete response (sCR), complete response (CR), and very good partial response (VGPR).
MRD negative | through study completion, up to 2 years
  MRD negative is defined as bone marrow MRD negative confirmed by new generation flow cytometry (NGF) or new generation sequencing technology (NGS) (the minimum detection sensitivity is that one clonal plasma cell can be detected from 105 nucleated cells);
continuous MRD negative rate | through study completion, up to 2 years
  Persistent MRD negative: new generation flow cytometry (NGF) or new generation sequencing technology (NGS) detects bone marrow MRD negative and imaging negative, with at least one year between two tests being negative
Overall survival (OS) | through study completion, up to 2 years
  Overall survival (OS) evaluation: defined as the time from enrollment to death.
Evaluation of duration of remission (DOR) | through study completion, up to 2 years
  Evaluation of duration of remission (DOR): defined as the time from the first response to treatment to disease progression or death

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Majithia N, Rajkumar SV, Lacy MQ, Buadi FK, Dispenzieri A, Gertz MA, Hayman SR, Dingli D, Kapoor P, Hwa L, Lust JA, Russell SJ, Go RS, Kyle RA, Kumar SK. Early relapse following initial therapy for multiple myeloma predicts poor outcomes in the era of novel agents. Leukemia. 2016 Nov;30(11):2208-2213. doi: 10.1038/leu.2016.147. Epub 2016 May 23. PMID 27211270
- [Background] Minnie SA, Hill GR. Immunotherapy of multiple myeloma. J Clin Invest. 2020 Apr 1;130(4):1565-1575. doi: 10.1172/JCI129205. PMID 32149732
- [Background] An G, Li Z, Tai YT, Acharya C, Li Q, Qin X, Yi S, Xu Y, Feng X, Li C, Zhao J, Shi L, Zang M, Deng S, Sui W, Hao M, Zou D, Zhao Y, Qi J, Cheng T, Ru K, Wang J, Anderson KC, Qiu L. The impact of clone size on the prognostic value of chromosome aberrations by fluorescence in situ hybridization in multiple myeloma. Clin Cancer Res. 2015 May 1;21(9):2148-56. doi: 10.1158/1078-0432.CCR-14-2576. Epub 2015 Feb 4. PMID 25652456
- [Background] An G, Acharya C, Feng X, Wen K, Zhong M, Zhang L, Munshi NC, Qiu L, Tai YT, Anderson KC. Osteoclasts promote immune suppressive microenvironment in multiple myeloma: therapeutic implication. Blood. 2016 Sep 22;128(12):1590-603. doi: 10.1182/blood-2016-03-707547. Epub 2016 Jul 14. PMID 27418644
- [Background] Riccardi A, Mora O, Tinelli C, Porta C, Danova M, Brugnatelli S, Grasso D, Tolca B, Spanedda R, De Paoli A, Barbarano L, Cavanna L, Giordano M, Delfini C, Nicoletti G, Bergonzi C, Rinaldi E, Piccinini L, Ascari E. Response to first-line chemotherapy and long-term survival in patients with multiple myeloma: results of the MM87 prospective randomised protocol. Eur J Cancer. 2003 Jan;39(1):31-7. doi: 10.1016/s0959-8049(02)00529-4. PMID 12504655
- [Background] Durie BG, Jacobson J, Barlogie B, Crowley J. Magnitude of response with myeloma frontline therapy does not predict outcome: importance of time to progression in southwest oncology group chemotherapy trials. J Clin Oncol. 2004 May 15;22(10):1857-63. doi: 10.1200/JCO.2004.05.111. Epub 2004 Apr 26. PMID 15111617
- [Background] Chinese Hematology Association; Chinese Society of Hematology. [Guidelines for the diagnosis and management of multiple myeloma in China (2022 revision)]. Zhonghua Nei Ke Za Zhi. 2022 May 1;61(5):480-487. doi: 10.3760/cma.j.cn112138-20220309-00165. Chinese. PMID 35488597
- [Background] Overdijk MB, Verploegen S, Bogels M, van Egmond M, Lammerts van Bueren JJ, Mutis T, Groen RW, Breij E, Martens AC, Bleeker WK, Parren PW. Antibody-mediated phagocytosis contributes to the anti-tumor activity of the therapeutic antibody daratumumab in lymphoma and multiple myeloma. MAbs. 2015;7(2):311-21. doi: 10.1080/19420862.2015.1007813. PMID 25760767
- [Background] Taylor RP, Lindorfer MA. Cytotoxic mechanisms of immunotherapy: Harnessing complement in the action of anti-tumor monoclonal antibodies. Semin Immunol. 2016 Jun;28(3):309-16. doi: 10.1016/j.smim.2016.03.003. Epub 2016 Mar 19. PMID 27009480
- [Background] Nijhof IS, Groen RW, Noort WA, van Kessel B, de Jong-Korlaar R, Bakker J, van Bueren JJ, Parren PW, Lokhorst HM, van de Donk NW, Martens AC, Mutis T. Preclinical Evidence for the Therapeutic Potential of CD38-Targeted Immuno-Chemotherapy in Multiple Myeloma Patients Refractory to Lenalidomide and Bortezomib. Clin Cancer Res. 2015 Jun 15;21(12):2802-10. doi: 10.1158/1078-0432.CCR-14-1813. Epub 2014 Nov 14. PMID 25398450
- [Background] Krejcik J, Casneuf T, Nijhof IS, Verbist B, Bald J, Plesner T, Syed K, Liu K, van de Donk NW, Weiss BM, Ahmadi T, Lokhorst HM, Mutis T, Sasser AK. Daratumumab depletes CD38+ immune regulatory cells, promotes T-cell expansion, and skews T-cell repertoire in multiple myeloma. Blood. 2016 Jul 21;128(3):384-94. doi: 10.1182/blood-2015-12-687749. Epub 2016 May 24. PMID 27222480
- [Background] van de Donk NWCJ, Usmani SZ. CD38 Antibodies in Multiple Myeloma: Mechanisms of Action and Modes of Resistance. Front Immunol. 2018 Sep 20;9:2134. doi: 10.3389/fimmu.2018.02134. eCollection 2018. PMID 30294326
- [Background] Voorhees PM, Kaufman JL, Laubach J, Sborov DW, Reeves B, Rodriguez C, Chari A, Silbermann R, Costa LJ, Anderson LD Jr, Nathwani N, Shah N, Efebera YA, Holstein SA, Costello C, Jakubowiak A, Wildes TM, Orlowski RZ, Shain KH, Cowan AJ, Murphy S, Lutska Y, Pei H, Ukropec J, Vermeulen J, de Boer C, Hoehn D, Lin TS, Richardson PG. Daratumumab, lenalidomide, bortezomib, and dexamethasone for transplant-eligible newly diagnosed multiple myeloma: the GRIFFIN trial. Blood. 2020 Aug 20;136(8):936-945. doi: 10.1182/blood.2020005288. PMID 32325490
- [Background] Palumbo A, Chanan-Khan A, Weisel K, Nooka AK, Masszi T, Beksac M, Spicka I, Hungria V, Munder M, Mateos MV, Mark TM, Qi M, Schecter J, Amin H, Qin X, Deraedt W, Ahmadi T, Spencer A, Sonneveld P; CASTOR Investigators. Daratumumab, Bortezomib, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Aug 25;375(8):754-66. doi: 10.1056/NEJMoa1606038. PMID 27557302
- [Background] McKeage K. Daratumumab: First Global Approval. Drugs. 2016 Feb;76(2):275-81. doi: 10.1007/s40265-015-0536-1. PMID 26729183
- [Background] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Background] Richardson PG, Oriol A, Beksac M, Liberati AM, Galli M, Schjesvold F, Lindsay J, Weisel K, White D, Facon T, San Miguel J, Sunami K, O'Gorman P, Sonneveld P, Robak P, Semochkin S, Schey S, Yu X, Doerr T, Bensmaine A, Biyukov T, Peluso T, Zaki M, Anderson K, Dimopoulos M; OPTIMISMM trial investigators. Pomalidomide, bortezomib, and dexamethasone for patients with relapsed or refractory multiple myeloma previously treated with lenalidomide (OPTIMISMM): a randomised, open-label, phase 3 trial. Lancet Oncol. 2019 Jun;20(6):781-794. doi: 10.1016/S1470-2045(19)30152-4. Epub 2019 May 13. PMID 31097405
- [Background] Cavo M, Gay F, Beksac M, Pantani L, Petrucci MT, Dimopoulos MA, Dozza L, van der Holt B, Zweegman S, Oliva S, van der Velden VHJ, Zamagni E, Palumbo GA, Patriarca F, Montefusco V, Galli M, Maisnar V, Gamberi B, Hansson M, Belotti A, Pour L, Ypma P, Grasso M, Croockewit A, Ballanti S, Offidani M, Vincelli ID, Zambello R, Liberati AM, Andersen NF, Broijl A, Troia R, Pascarella A, Benevolo G, Levin MD, Bos G, Ludwig H, Aquino S, Morelli AM, Wu KL, Boersma R, Hajek R, Durian M, von dem Borne PA, Caravita di Toritto T, Zander T, Driessen C, Specchia G, Waage A, Gimsing P, Mellqvist UH, van Marwijk Kooy M, Minnema M, Mandigers C, Cafro AM, Palmas A, Carvalho S, Spencer A, Boccadoro M, Sonneveld P. Autologous haematopoietic stem-cell transplantation versus bortezomib-melphalan-prednisone, with or without bortezomib-lenalidomide-dexamethasone consolidation therapy, and lenalidomide maintenance for newly diagnosed multiple myeloma (EMN02/HO95): a multicentre, randomised, open-label, phase 3 study. Lancet Haematol. 2020 Jun;7(6):e456-e468. doi: 10.1016/S2352-3026(20)30099-5. Epub 2020 Apr 30. PMID 32359506
- [Background] van der Veer MS, de Weers M, van Kessel B, Bakker JM, Wittebol S, Parren PW, Lokhorst HM, Mutis T. Towards effective immunotherapy of myeloma: enhanced elimination of myeloma cells by combination of lenalidomide with the human CD38 monoclonal antibody daratumumab. Haematologica. 2011 Feb;96(2):284-90. doi: 10.3324/haematol.2010.030759. Epub 2010 Nov 25. PMID 21109694
- [Background] Sehgal K, Das R, Zhang L, Verma R, Deng Y, Kocoglu M, Vasquez J, Koduru S, Ren Y, Wang M, Couto S, Breider M, Hansel D, Seropian S, Cooper D, Thakurta A, Yao X, Dhodapkar KM, Dhodapkar MV. Clinical and pharmacodynamic analysis of pomalidomide dosing strategies in myeloma: impact of immune activation and cereblon targets. Blood. 2015 Jun 25;125(26):4042-51. doi: 10.1182/blood-2014-11-611426. Epub 2015 Apr 13. PMID 25869284
- [Background] Dimopoulos MA, Terpos E, Boccadoro M, Delimpasi S, Beksac M, Katodritou E, Moreau P, Baldini L, Symeonidis A, Bila J, Oriol A, Mateos MV, Einsele H, Orfanidis I, Ahmadi T, Ukropec J, Kampfenkel T, Schecter JM, Qiu Y, Amin H, Vermeulen J, Carson R, Sonneveld P; APOLLO Trial Investigators. Daratumumab plus pomalidomide and dexamethasone versus pomalidomide and dexamethasone alone in previously treated multiple myeloma (APOLLO): an open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Jun;22(6):801-812. doi: 10.1016/S1470-2045(21)00128-5. PMID 34087126
- [Background] Chari A, Suvannasankha A, Fay JW, Arnulf B, Kaufman JL, Ifthikharuddin JJ, Weiss BM, Krishnan A, Lentzsch S, Comenzo R, Wang J, Nottage K, Chiu C, Khokhar NZ, Ahmadi T, Lonial S. Daratumumab plus pomalidomide and dexamethasone in relapsed and/or refractory multiple myeloma. Blood. 2017 Aug 24;130(8):974-981. doi: 10.1182/blood-2017-05-785246. Epub 2017 Jun 21. PMID 28637662
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Background] Larocca A, Dold SM, Zweegman S, Terpos E, Wasch R, D'Agostino M, Scheubeck S, Goldschmidt H, Gay F, Cavo M, Ludwig H, Straka C, Bringhen S, Auner HW, Caers J, Gramatzki M, Offidani M, Dimopoulos MA, Einsele H, Boccadoro M, Sonneveld P, Engelhardt M. Patient-centered practice in elderly myeloma patients: an overview and consensus from the European Myeloma Network (EMN). Leukemia. 2018 Aug;32(8):1697-1712. doi: 10.1038/s41375-018-0142-9. Epub 2018 Apr 25. PMID 29880892
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Background] Rajkumar SV, Harousseau JL, Durie B, Anderson KC, Dimopoulos M, Kyle R, Blade J, Richardson P, Orlowski R, Siegel D, Jagannath S, Facon T, Avet-Loiseau H, Lonial S, Palumbo A, Zonder J, Ludwig H, Vesole D, Sezer O, Munshi NC, San Miguel J; International Myeloma Workshop Consensus Panel 1. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011 May 5;117(18):4691-5. doi: 10.1182/blood-2010-10-299487. Epub 2011 Feb 3. PMID 21292775
- [Background] Callander NS, Baljevic M, Adekola K, Anderson LD, Campagnaro E, Castillo JJ, Costello C, Devarakonda S, Elsedawy N, Faiman M, Garfall A, Godby K, Hillengass J, Holmberg L, Htut M, Huff CA, Hultcrantz M, Kang Y, Larson S, Liedtke M, Martin T, Omel J, Sborov D, Shain K, Stockerl-Goldstein K, Weber D, Berardi RA, Kumar R, Kumar SK. NCCN Guidelines(R) Insights: Multiple Myeloma, Version 3.2022. J Natl Compr Canc Netw. 2022 Jan;20(1):8-19. doi: 10.6004/jnccn.2022.0002. PMID 34991075